CLINICAL TRIAL: NCT03122288
Title: Individualized-Targeted Cognitive Training in Older Adults With HAND
Brief Title: Individualized Cognitive Training in HIV
Acronym: TOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, David Vance, PhD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F161122002; 1R21NR016632-01 (NIH)
Record Dates: First submitted 2017-04-11; First posted 2017-04-20 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: HIV-Associated Cognitive Motor Complex; Aging; Cognitive Impairment; Cognitive Decline; Attention Impaired; Processing, Visual Spatial; Cognitive Deficit in Attention; Cognitive Disorder in Remission
MeSH Terms: conditions — AIDS Dementia Complex; Cognitive Dysfunction; Spatial Processing | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A pre-post two-group experimental design will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Cognitive Training (Experimental): Participants randomized to this arm will receive 20 hours of computerized cognitive training in the two predominate cognitive domains in which they experience deficits that contribute to their HIV-Associated Neurocognitive Disorder diagnosis.
  Interventions: Behavioral: Individualized Cognitive Training
- No-Contact Control (Other): Participants in this arm will not receive any experimental or sham contact. They will only participate in the Baseline and Posttest assessments.
  Interventions: Other: No-Contact Control

INTERVENTIONS:
Behavioral: Individualized Cognitive Training — These are specific computerized exercises that are designed to improve performance in particular cognitive domains (e.g., attention, speed of processing, verbal learning/memory).
  Other Names: Insight Software
  Arms: Individualized Cognitive Training
Other: No-Contact Control — This is simply a no-contact control group. Participants in this group will receive no additional contact with the study beyond the baseline and posttest assessments.
  Other Names: Control Group
  Arms: No-Contact Control

SUMMARY:
Over 50% of adults with HIV have some form of HIV-Associated Neurocognitive Disorder (HAND) which represents a significant symptom that interferes with everyday functioning and quality of life. As adults age with HIV, they are more likely to develop comorbidities such as cardiovascular disease, hypertension, and insulin resistance which will further contribute to poorer cognitive functioning and HAND. Based upon the Frascati criteria, HAND is diagnosed when a person performs less than 1 to 2 SD below their normative mean (education & age) on measures of two or more cognitive domains (e.g., attention, speed of processing, verbal memory, executive functioning). Yet, from the cognitive literature and prior studies, administering certain computerized cognitive training programs may improve specific cognitive domains in older adults and those with HIV. Such cognitive training programs may be effective in older adults with HIV and therefore investigators may be able to change the diagnosis of HAND in such cognitively vulnerable adults. In this pre-post experimental study, 146 older adults (50+) with HAND will be randomized to be in either: 1) the Individualied-Targeted Cognitive Training, or 2) a no-contact control group. The investigators will focus on those cognitive domains in which participants express an impairment and train them with the corresponding cognitive program. Such an Individualized-Targeted Cognitive Training approach using standard cognitive training programs may offer hope and symptom relief to those individuals diagnosed with HAND. Furthermore, these changes may result in improved everyday functioning (e.g., IADLs) and quality of life. This approach represents a paradigm shift in possibly changing the way HAND is examined. Specific Aim 1: Compare adults who do receive Individualized-Targeted Cognitive Training to those who do not in order to determine whether a change in HAND prevalence and severity occurs between groups. Exploratory Aim 1: Compare adults who do receive individualized-targeted cognitive training to those who do not in order to determine whether this improves everyday functioning (e.g., IADLs). Exploratory Aim 2: Determine whether improvements in HAND and/or everyday functioning over time mediate improvements in quality of life.

DETAILED DESCRIPTION:
This research directly meets the goals of the NIH Cognitive and Emotional Health Project and the Healthy Brain Initiative which seek to "maintain or improve the cognitive performance of all adults," especially for "populations experiencing the greatest disparities and risks in cognitive health."

Significance: Using the Frascati criteria, 52% - 59% of people with HIV experience some form of HIV-Associated Neurocognitive Disorder (HAND) which affects medication adherence, instrumental activities of daily living (IADLs), and even mood maintenance and quality of life. By 2020, 70% of adults with HIV in the United States will be 50 and older; thus, cognitive aging in this group represents a major concern. In a prior study (R03MH076642-01A2) conducted in the HAART era, when comparing cognitive functioning between older and younger HIV-positive and HIV-negative adults, older adults with HIV performed the worst. In the HAART era, these cognitive impairments continue to be observed in several cognitive domains including memory, learning, executive functioning, and speed of processing.

Regrettably, few behavioral interventions aimed at improving cognition in this pharmacologically-burdened population have been attempted. Pharmacological interventions have short-lived effects, if any, and can produce adverse side effects in a population prone to multiple comorbidities. Fortunately, computerized cognitive training interventions have been shown to improve cognition without adverse side-effects. Yet, only two types of computerized cognitive training interventions have been studied in adults with HIV. Becker and colleagues partially randomized 60 adults with HIV and without HIV to engage in 14 computerized targeted modules (e.g., knowledge, memory) over 24 weeks. No significant effects were found; however, adherence was poor. In a prior study, investigators randomized 46 adults to either a speed of processing training (10 hrs of training) group or a no-contact control group. Adherence was excellent and improvements were observed on this cognitive domain which transferred to an everyday functioning task.

Despite this lack of cognitive training studies in HIV, studies in older adults have shown their efficacy in improving specific cognitive abilities, some as much as 1-1.5 standard deviations (SD) above baseline performance or age/education-based norms. Using Frascati criteria, HAND is diagnosed when a person performs at least 1 to 2 SD below their normative mean on measures of two or more cognitive domains (e.g., verbal memory, speed of processing, executive functioning); yet many individuals may be only a fraction of a SD below the cut off. A meta-analysis of 52 cognitive training studies indicated the average cognitive improvement following cognitive training was 0.22 SD. Although this seems to be a small to moderate effect size, such cognitive training programs can change the diagnosis of HAND for some by improving cognitive performance to within acceptable performance norms. In this study, older adults (50+) with HAND will be enrolled to determine which cognitive domains are attributable to their diagnosis. Then those cognitive domains in which they have impairments will be targeted for training with the corresponding cognitive program. Such a tailored approach to standard cognitive training programs may offer hope and symptom relief to those individuals diagnosed with HAND. Furthermore, these changes may result in improved everyday functioning and quality of life. This approach also represents a paradigm shift in changing the way clinicians and researchers look at HAND in that this is not a static "progressive" diagnosis; Antinori et al. observed a 20% fluctuation of HAND over as little as 1 year, with some improving or declining in their cognitive performance. Such fluctuations, at least partially, reflect positive neuroplasticity that can be manipulated with cognitive training to improve cognition which can improve medication adherence and other IADLs. This study will use a basic two group pre-post experimental design of 146 adults with HAND.

ELIGIBILITY:
Inclusion Criteria:

* Must be 40+ years
* English speaking
* Have HIV-Associated Neurocognitive Disorder (HAND)

Exclusion Criteria:

* Because the study requires several weeks, participants not living in stable housing (e.g., halfway house) will be excluded.
* Participants with significant neuromedical co-morbidities (e.g., schizophrenia, epilepsy, bipolar disorder, multiple sclerosis, Alzheimer's disease or related dementias, mental retardation)
* Currently undergoing radiation or chemotherapy
* A history of brain trauma with a loss of consciousness greater than 30 minutes
* Legally blind or deaf

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Prevalence and Severity of HIV-Associated Neurocognitive Disorder (HAND) as Measured by Neurocognitive Tests Interpreted by the Frascati Criteria | Per participants, approximately 10-12 weeks
  Compare adults who do receive Individualized-Targeted Cognitive Training to those who do not in order to determine whether a change in HAND prevalence and severity occurs between groups. A battery of neurocognitive tests (e.g., Trails Making Test A, Trails Making Test B, etc.) of different domains (e.g., speed of processing, verbal memory, etc.) are used which are normed by age/education which are then use with the Frascati Criteria (a neurological algorithm to classify cognitive impairment) to determine HIV-Associated Neurocognitive Disorder, both presence and severity (i.e., Global Severity Rating). This is administered at baseline and posttest.

SECONDARY OUTCOMES:
Improvement on Everyday Functioning as Measured by the Timed Instrumental Activities of Daily Living Test | Per participants, approximately 10-12 weeks
  The Timed Instrumental Activities of Daily Living Test -- This test measures the accuracy and time it takes to perform 5 IADLs (e.g., counting out correct change, reading ingredients on a can of food). Slower speed of processing is associated with longer times to complete these tasks, even after adjusting for age, education level, depression, and general health. The time from each of the 5 IADLs is added together to form a composite score. Test-retest reliability is 0.64. This test is administered at baseline and posttest.
Improvement on Everyday Functioning as Measured by the Medication Adherence Scale | Per participants, approximately 10-12 weeks
  Medication Adherence - This IADL is measured by the Simplified Medication Adherence Questionnaire (as well as virological control). It consists of sixl items that ask about how consistently one takes his/her medications; the items can be summed to form a composite score. This measure is validated with virological outcomes and has good internal consistency (α = 0.75) and inter-observer agreement (88.2%). This questionnaire is administered at baseline and posttest.
Improvement in Quality of Life as Measured by Depression | Per participants, approximately 10-12 weeks
  Centers for Epidemiological Studies - Depression Scale (CES-D) - This depression scale measures how often (not at all - extremely) participants acknowledge 20 verbal symptoms of depression; score are tallied to form a composite score; higher scores indicate greater self-reported depressive symptomatology. Cronbach's α is very good at 0.88. This scale is administered at baseline and posttest.
Improvement in Quality of Life as Measured by Internal Locus of Control | Per participants, approximately 10-12 weeks
  Internal Locus of Control - This six (6-point Likert-type) item measure assesses the degree to which participants perceive that they can exert influence over their life. The items are summed to form a composite score; higher scores indicate more internal locus of control. Cronbach's α's range from 0.62 to 0.79. This measure is administered at baseline and posttest.
Improvement in Quality of Life as Measured by Health-Related Quality of Life | Per participants, approximately 10-12 weeks
  Medical Outcomes Study Short Form (SF-36)/Health-Related Quality of Life - SF-36 assesses health-related quality of life which is a subscale of this measure. The item of this subscale are summed to form a composite score. In the ACTIVE Study, improvement on this variable was observed in the speed of processing training group. Cronbach's α is greater than 0.85. This subscale is administered at baseline and posttest.
Improvement in Quality of Life as Measured by Self-Rated Health | Per participants, approximately 10-12 weeks
  Medical Outcomes Study Short Form (SF-36)/Self-Rated Health - SF-36 assesses self-rated health on only 1 item which is a Likert type scale (In general, I would say that my health is: Excellent, Very Good, Good, Fair, Poor). In the ACTIVE Study, improvement on self-rated health was observed in the speed of processing training group. This item is administered at baseline and posttest.
Improvement in Quality of Life as Measured by Cognitive Complaints | Per participants, approximately 10-12 weeks
  Cognitive Failures Questionnaire (CFQ) - CFQ assesses common everyday cognitive complaints one may have such as in memory (e.g., "Do you forget where you put something like a newspaper or book?"). All of the 25 items on this measure are summed to form an overall composite score; higher scores are indicative of greater subjective cognitive complaints. This questionnaire is administered at baseline and posttest.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vance DE, Fazeli PL, Ross LA, Wadley VG, Ball KK. Speed of processing training with middle-age and older adults with HIV: a pilot study. J Assoc Nurses AIDS Care. 2012 Nov-Dec;23(6):500-10. doi: 10.1016/j.jana.2012.01.005. Epub 2012 May 11. PMID 22579081
- [Background] Vance DE, Fazeli PL, Moneyham L, Keltner NL, Raper JL. Assessing and treating forgetfulness and cognitive problems in adults with HIV. J Assoc Nurses AIDS Care. 2013 Jan-Feb;24(1 Suppl):S40-60. doi: 10.1016/j.jana.2012.03.006. PMID 23290376
- [Background] Vance DE. Prevention, Rehabilitation, and Mitigation Strategies of Cognitive Deficits in Aging with HIV: Implications for Practice and Research. ISRN Nurs. 2013;2013:297173. doi: 10.1155/2013/297173. Epub 2013 Feb 3. PMID 23431469
- [Background] Lin F, Chen DG, Vance D, Mapstone M. Trajectories of combined laboratory- and real world-based speed of processing in community-dwelling older adults. J Gerontol B Psychol Sci Soc Sci. 2013 May;68(3):364-73. doi: 10.1093/geronb/gbs075. Epub 2012 Sep 11. PMID 22967505
- [Background] Fazeli PL, Ross LA, Vance DE, Ball K. The relationship between computer experience and computerized cognitive test performance among older adults. J Gerontol B Psychol Sci Soc Sci. 2013 May;68(3):337-46. doi: 10.1093/geronb/gbs071. Epub 2012 Aug 28. PMID 22929395
- [Background] Kaur J, Dodson JE, Steadman L, Vance DE. Predictors of improvement following speed of processing training in middle-aged and older adults with HIV: a pilot study. J Neurosci Nurs. 2014 Feb;46(1):23-33. doi: 10.1097/JNN.0000000000000034. PMID 24399164
- [Derived] Byun JY, Azuero A, Fazeli PL, Li W, Chapman Lambert C, Del Bene VA, Triebel K, Jacob A, Vance DE. Perceived Improvement and Satisfaction With Training After Individualized-Targeted Computerized Cognitive Training in Adults With HIV-Associated Neurocognitive Disorder Living in Alabama: A Descriptive Cross-sectional Study. J Assoc Nurses AIDS Care. 2022 Sep-Oct 01;33(5):581-586. doi: 10.1097/JNC.0000000000000333. Epub 2022 Apr 1. No abstract available. PMID 35363623
- [Derived] Vance DE, Pope CN, Fazeli PL, Azuero A, Frank JS, Wadley VG, Raper JL, Byun JY, Ball KK. A Randomized Clinical Trial on the Impact of Individually Targeted Computerized Cognitive Training on Quality of Life Indicators in Adults With HIV-Associated Neurocognitive Disorder in the Southeastern United States. J Assoc Nurses AIDS Care. 2022 May-Jun 01;33(3):295-310. doi: 10.1097/JNC.0000000000000316. Epub 2021 Dec 6. PMID 34864757
- [Derived] Waldrop D, Irwin C, Nicholson WC, Lee CA, Webel A, Fazeli PL, Vance DE. The Intersection of Cognitive Ability and HIV: A Review of the State of the Nursing Science. J Assoc Nurses AIDS Care. 2021 May-Jun 01;32(3):306-321. doi: 10.1097/JNC.0000000000000232. PMID 33449578
- [Derived] Vance DE, Robinson J, Walker TJ, Tende F, Bradley B, Diehl D, McKie P, Fazeli PL. Reactions to a Probable Diagnosis of HIV-Associated Neurocognitive Disorder: A Content Analysis. J Assoc Nurses AIDS Care. 2020 May-Jun;31(3):279-289. doi: 10.1097/JNC.0000000000000120. PMID 31436599
- [Derived] Vance DE, Cody SL, Nicholson WC, Cheatwood J, Morrison S, Fazeli PL. The Association Between Olfactory Function and Cognition in Aging African American and Caucasian Men With HIV: A Pilot Study. J Assoc Nurses AIDS Care. 2019 Sep-Oct;30(5):e144-e155. doi: 10.1097/JNC.0000000000000086. PMID 31259847
- [Derived] Vance DE, Lee L, Munoz-Moreno JA, Morrison S, Overton T, Willig A, Fazeli PL. Cognitive Reserve Over the Lifespan: Neurocognitive Implications for Aging With HIV. J Assoc Nurses AIDS Care. 2019 Sep-Oct;30(5):e109-e121. doi: 10.1097/JNC.0000000000000071. PMID 30865059
- [Derived] Vance DE, Cody SL, Nicholson C, Cheatwood J, Morrison S, Fazeli PL. Olfactory Dysfunction in Aging African American and Caucasian Men With HIV: A Pilot Study. J Assoc Nurses AIDS Care. 2022 May-Jun 01;33(3):e19-e30. doi: 10.1097/JNC.0000000000000061. PMID 30676359
- [Derived] Vance DE, Fazeli PL, Cheatwood J, Nicholson WC, Morrison SA, Moneyham LD. Computerized Cognitive Training for the Neurocognitive Complications of HIV Infection: A Systematic Review. J Assoc Nurses AIDS Care. 2019 Jan-Feb;30(1):51-72. doi: 10.1097/JNC.0000000000000030. PMID 30586083
- [Derived] Vance DE, Blake BJ, Brennan-Ing M, DeMarco RF, Fazeli PL, Relf MV. Revisiting Successful Aging With HIV Through a Revised Biopsychosocial Model: An Update of the Literature. J Assoc Nurses AIDS Care. 2019 Jan-Feb;30(1):5-14. doi: 10.1097/JNC.0000000000000029. PMID 30586079
- [Derived] Vance DE, Jensen M, Tende F, Raper JL, Morrison S, Fazeli PL. Individualized-Targeted Computerized Cognitive Training to Treat HIV-Associated Neurocognitive Disorder: An Interim Descriptive Analysis. J Assoc Nurses AIDS Care. 2018 Jul-Aug;29(4):604-611. doi: 10.1016/j.jana.2018.04.005. Epub 2018 Apr 23. No abstract available. PMID 29764716